CLINICAL TRIAL: NCT02269813
Title: PRospective Study to Measure the Impact of MammaPrint on Adjuvant Treatment in Hormone Receptor-positive HER2-negative Breast Cancer Patients (PRIMe)
Acronym: PRIMe
Status: Completed | Type: Observational
Sponsor: West German Study Group (Other)
Collaborators: Agendia (Industry)
Responsible Party: Sponsor
Other Study IDs: WSG-PRIMe
Record Dates: First submitted 2014-10-14; First posted 2014-10-21 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer
Keywords: MammaPrint; BluePrint; TargetPrint
MeSH Terms: conditions — Breast Neoplasms | interventions — Blueprint Asept

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ET/GOOD: Endocrine therapy only.
  Interventions: Other: MammaPrint; Other: BluePrint; Other: TargetPrint
- CT/POOR: Chemoendocrine therapy according to national guidelines.
  Interventions: Other: MammaPrint; Other: BluePrint; Other: TargetPrint

INTERVENTIONS:
Other: MammaPrint
Other: BluePrint
Other: TargetPrint

SUMMARY:
PRIMe is a prospective, case-only trial designed to measure the impact of MammaPrint on physician chemotherapy intention in the two discordant groups (ET/POOR, CT/GOOD) in stage 1 and 2 HR-positive HER2-negative breast cancer patients. The design also provides for assessment of several important secondary indicators. Eligible patients will have their tumor sample analyzed for MammaPrint, BluePrint and TargetPrint. Patients cannot start treatment before the MammaPrint result is received and taken into consideration for the adjuvant treatment plan.

ELIGIBILITY:
Inclusion Criteria:

* Women with histologically proven invasive stage 1 and 2 breast cancer
* Hormone receptor positive according to local standards
* HER2 negative - i.e. IHC 0-1+, or FISH or other ISH non-amplified (locally assessed)
* Axillary lymph node status: 0-3 involved (macro metastases i.e. >2mm OR micro metastases i.e. >0.2-2mm)
* ≥ 18 years of age at time of consent
* Patients must be eligible to receive adjuvant chemotherapy and endocrine therapy as defined by a good Karnofsky index, no hematological, cardiological or hepatic contraindications nor any impeding comorbidity
* Written informed consent

Exclusion Criteria:

* ≥4 involved axillary nodes
* Multi-centric disease with more than 2 clinically relevant lesions
* HR negative OR HER2 positive/amplified (locally assessed)
* Previous diagnosis of malignancy unless disease free for 10 years
* Metastatic disease
* Tumor sample shipped to Agendia with ≤ 30% tumor cells or that fails QA or QC criteria
* Women who have started or completed adjuvant chemotherapy or neo-adjuvant chemotherapy for current breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will comprise patients for whom the investigator will advise either endocrine therapy or chemotherapy + endocrine therapy. Patients confirmed to be low/high risk by the gene signature will receive the respective treatment. Patients with discordant results will be investigated for investigator's chemotherapy intention after MammaPrint results are available.
Sampling Method: Probability Sample
Enrollment: 452 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Measure the impact of MammaPrint on adjuvant treatment decisions in discordant groups (ET/POOR and CT/GOOD) in stage-1/2, HR+, HER2- breast cancer and test whether these impacts each exceed a pre-determined compliance threshold. | Up to 6 months after end of treatment.
  Compliance, assessed in terms of the fraction of patients in each discordant group whose physicians switch their chemotherapy intention following MammaPrint test disclosure is used to measure the impact of MammaPrint on adjuvant treatment decisions.
Assess the incremental cost-effectiveness of MammaPrint in terms of cost and quality-adjusted life years within a health economic context using the impacts measured in this trial as well as the predictive impact demonstrated in previous trials. | Up to 6 months after end of treatment.

SECONDARY OUTCOMES:
Measure the impacts of MammaPrint on adjuvant treatment decisions (physician chemotherapy intention) and compare with previous trials involving MammaPrint or other tests. | Up to 6 months after end of treatment.
  The planned analysis includes assessment of the incremental cost-effectiveness (ICER) of MammaPrint within a health economic context (i.e., taking cost and quality-adjusted life years into account).
Measure rate (by incidence) and severity (by Common Toxicity Criteria) of treatment-related serious adverse events stratified by whether or not patient received adjuvant chemotherapy. | Up to 6 months after end of treatment.
Assess change in patients' decisional conflict status and anxiety levels before and after MammaPrint results via questionnaire, stratified by the four groups (2 concordant and 2 discordant). | Up to 6 months after end of treatment.
Assess investigators' confidence in treatment recommendations before and after MammaPrint results were known via questionnaire. | Up to 6 months after end of treatment.
Assess concordance of final treatment intention and treatment actually received by number of patients. | Up to 6 months after end of treatment.
Assess concordance of TargetPrint ER, PR and HER2 results with locally assessed IHC/FISH ER, PR and HER2 by number of patients. | Up to 6 months after end of treatment.
Compare clinical subtype based on IHC/FISH ER, PR, HER2 and Ki-67 (St Gallen 2013) with BluePrint molecular subtype by diagnostic definition of subtype. | Up to 6 months after end of treatment.
Assess concordance of MammaPrint, BluePrint and TargetPrint in multi-centric breast cancer by number of patients. | Up to 6 months after end of treatment.
Assess the combined switch rate in the two concordant groups (ET/GOOD) and (CT/POOR) and verify that it is lower than the switch rate in both discordant groups by number of patients. | Up to 6 months after end of treatment.
Perform descriptive sub-analysis in pre- and post-menopausal women by switch percentages. | Up to 6 months after end of treatment.
Perform cross-validation with other adjuvant breast cancer studies by switch rate, if available. | Up to 6 months after end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Harbeck, Prof. Dr., Principal Investigator — Scientific Director; Ulrike Nitz, Prof. Dr., Study Chair — General Manager/Medical Director
Locations (3):
- Medizinische Universität Innsbruck Universitätsklinik für Frauenheilkunde, Innsbruck, Austria
- Breast Center of the University of Munich (LMU), Munich, Germany
- Kantonsspital St.Gallen, Sankt Gallen, Switzerland